### Janssen Research & Development

### **Statistical Analysis Plan**

A Randomized, Double-blind, Event-driven, Placebo-controlled, Multicenter Study of the Effects of Canagliflozin on Renal and Cardiovascular Outcomes in Subjects With Type 2 Diabetes Mellitus and Diabetic Nephropathy

**Protocol 28431754DNE3001; Phase 3** 

JNJ-28431754 (canagliflozin)

**Amendment 2** 

Status: Approved
Date: 1 June 2018

Prepared by: Janssen Research & Development, LLC

Document No.: EDMS-ERI-85306295, 2.0

Compliance: The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TABL | BLE OF CONTENTS2 | |
|---|---|---|
| ABBR | REVIATIONS | 4 |
| 1. I | INTRODUCTION | 6 |
| 1.1. | Trial Objectives | |
| 1.2. | Trial Design | |
| 1.3. | Statistical Hypothesis for Trial Objectives | |
| 1.4. | Sample Size Justification | |
| 1.5. | Randomization, Blinding, and Stratification | 9 |
| 2. ( | GENERAL ANALYSIS DEFINITIONS | 10 |
| 2.1. | Analysis Populations | |
| 2.2. | Analysis Sets | 10 |
| 2.3. | Time-to-Event Data | 10 |
| 2.3.1. | Subject-Level Trial Milestone Dates | 10 |
| 2.3.2. | Censoring Rules | 12 |
| 2.4. | Visit Windows | 12 |
| 3. I | INTERIM ANALYSIS | 13 |
| 4. \$ | SUBJECT INFORMATION | 14 |
| 4.1. | Baseline Anthropometric and Demographic Characteristics | |
| 4.1.1. | Baseline Disease Characteristics | |
| 4.2. | Disposition Information | |
| 4.3. | Extent of Exposure and Follow-Up | |
| 4.4. | Prior and Concomitant Medications | |
| 4.5. | Patient Management of Cardiovascular Risk Factors | |
| | EFFICACY | 17 |
| 5.1.1. | Level of Significance | 17 |
| 5.1.2. | Data Handling Rules | 17 |
| 5.2. | Primary Efficacy Endpoint | 18 |
| 5.2.1. | Definition | 18 |
| 5.2.2. | , | |
| 5.2.2.1 | - 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
| 5.2.2.1 | and the second s | |
| 5.3. | Subgroup Analyses for the Primary Endpoint | |
| 5.4. | Major Secondary Endpoints | |
| 5.4.1. | Definition | |
| 5.4.2. | Analysis Methods | |
| 5.5. | Multiplicity Adjustment | |
| 5.6. | Other Efficacy Analyses | |
| 5.6.1. | Definition of Exploratory Efficacy Endpoints | |
| 5.6.2. | Definition of Other Efficacy Endpoints | |
| 5.6.3. | Analysis Methods for Other Efficacy Analyses | 23 |
| | SAFETY | |
| 6.1. | Adverse Events | |
| 6.1.1. | General Adverse Events | |
| 6.2. | Adverse Events of Interest | |
| 6.3. | Modified Rankin Scores for Stroke | |
| 6.4. | Hypoglycemia | 27 |

# Statistical Analysis Plan 28431754DNE3001; Phase 3

| 6.5. | Clinical Laboratory Tests | 28 |
|---|---|---|
| 6.6. | Vital Signs | 29 |
| REFI | ERENCES | 30 |
| ATT | ACHMENT 1 | 31 |
| 1. | DIURETICS | 32 |
| | Diuretics [loop] | |
| 1.2. | Diuretics [non-loop] | |
| ATT | ACHMENT 2 | 39 |
| 1. | MEDICAL HISTORY | 39 |
| 1.1. | Hypertension | |
| 1.2. | Dyslipidemia | |
| 1.3. | Fractures | |
| 2. | LIST OF PREFERRED TERMS FOR SELECTED ADVERSE EVENTS OF INTEREST | <b>4</b> 1 |
| ATT | ACHMENT 3 | 51 |
| CLIN | IICAL LABORATORY TESTS | 51 |
| ATT | ACHMENT 4 | 52 |
| CRIT | ERIA FOR PRE-DEFINED LIMIT OF CHANGE (PDLC) AND ABNORMAL VALUES | 52 |

#### **ABBREVIATIONS**

ACEi angiotensin-converting enzyme inhibitor

AE adverse event

AHA antihyperglycemic agent
ARB angiotensin-receptor blockers
ATC Anatomical Therapeutic Chemical

BMI body mass index
CI confidence interval
CKD chronic kidney disease
CM concomitant medication

CV cardiovascular

DBP diastolic blood pressure

eGFR estimated glomerular filtration rate

ESKD end-stage kidney disease
GCP Good Clinical Practice
GTED global trial end date
HbA<sub>1c</sub> hemoglobin A<sub>1c</sub>

HDL-C high-density lipoprotein cholesterol

IEAC Independent Endpoint Adjudication Committee

IWRS Interactive Web Response System LDL-C low-density lipoprotein cholesterol

MH medical history

MedDRA Medical Dictionary for Regulatory Activities

ITT intent-to-treat

MACE major adverse cardiovascular event

MI myocardial infarction
PDLC pre-defined limit of change

QD once daily
ROW Rest of the World
SAP statistical analysis plan
SBP systolic blood pressure
SD standard deviation

SGLT2 sodium-glucose co-transporter 2 SMBG self-monitored blood glucose

SI standard units
SOC system organ class
T2DM type 2 diabetes mellitus
TEAE treatment-emergent AE
UACR urinary albumin/creatinine ratio
UILN upper limit of normal

VS vital sign

WHODRUG World Health Organization Drug Utilization Research Group

#### Amendment 1 (September 11, 2017)

The major changes in this amendment include the clarification of alpha spending in the interim and the final analysis, the decrease of the number of primary composite events required for the interim analysis from 420 to 405, and re-ordering of the secondary endpoints as well as the addition of 2 new endpoints (MACE and hospitalized congestive heart failure) in the list of secondary endpoints.

#### Amendment 2 (June 1, 2018)

The reason for this amendment is to update the alpha level used for testing the secondary efficacy endpoints and include other minor clarifications of the analyses.

Approved, Date: 1 June 2018

#### 1. INTRODUCTION

This statistical analysis plan (SAP) contains the definitions of analysis sets, derived variables, and statistical methods for the final analyses of efficacy and safety data from the canagliflozin study 28431754DNE3001. An interim analysis will be conducted when the mean duration of follow-up is at least 2 years and the events within the primary composite have been adjudicated as endpoints in approximately 405 subjects. Details regarding the interim analysis will be provided in a separate SAP.

# 1.1. Trial Objectives

### **Primary Objective**

In subjects with type 2 diabetes mellitus (T2DM), Stage 2 or 3 chronic kidney disease (CKD) and macroalbuminuria who are receiving standard of care, to assess the efficacy of canagliflozin relative to placebo in reducing:

• the composite endpoint of end-stage kidney disease (ESKD), doubling of serum creatinine, and renal or cardiovascular (CV) death.

## **Secondary Objectives**

In subjects with T2DM, Stage 2 or 3 CKD and macroalbuminuria who are receiving standard of care, to assess the efficacy of canagliflozin relative to placebo in reducing:

- the composite endpoint of CV death and hospitalized congestive heart failure
- the composite endpoint of CV death, non-fatal myocardial infarction (MI), and non-fatal stroke (ie, 3-point major adverse cardiac event [MACE])
- hospitalized congestive heart failure
- the renal composite endpoint of ESKD, doubling of serum creatinine, and renal death
- CV death
- all-cause death
- the CV composite endpoint of CV death, non-fatal MI, non-fatal stroke, hospitalized congestive heart failure, and hospitalized unstable angina

### **Exploratory Objectives**

In subjects with T2DM, Stage 2 or 3 CKD and macroalbuminuria who are receiving standard of care, to assess efficacy of canagliflozin relative to placebo in reducing:

• the composite endpoint of ESKD, renal or CV death

• individual components of the renal and cardiovascular composite endpoints (ESKD, doubling of serum creatinine, renal death, CV death, fatal or non-fatal MI, fatal or non-fatal stroke, hospitalized congestive heart failure, hospitalized unstable angina)

and to assess the impact of canagliflozin relative to placebo on:

- changes in estimated glomerular filtration rate (eGFR) over time
- changes in urinary albumin-to-creatinine ratio (UACR) over time

# **Safety Objective**

To assess the overall safety and tolerability of canagliflozin.

## 1.2. Trial Design

This is a randomized, double-blind, placebo-controlled, parallel-group, 2-arm, multicenter study that will include a total of approximately 4,200 subjects. The study will have a pretreatment phase, consisting of a prescreening, screening (up to 8 weeks), and 2-week single-blind placebo run-in phase. Subjects will be prescreened on the basis of eGFR and UACR. Only subjects with an eGFR of  $\geq$ 30 to  $\leq$ 90 mL/min/1.73m² and a UACR of level  $\geq$ 300 mg/g to  $\leq$ 5,000 mg/g (as confirmed by a local laboratory within the 3 months prior to screening) will be eligible for screening by the central laboratory.

Subjects must be on a maximum tolerated labeled daily dose of an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) for a period of at least 4 weeks prior to randomization. To reach this requirement, the screening phase may be extended (up to 8 weeks). In addition, other anti-hypertensive, lipid-lowering and antihyperglycemic therapies should also be dose stable prior to randomization.

Subjects who meet all entry criteria will enter the single-blind placebo run-in phase at Week -2. During this phase, subjects will be instructed to take one capsule daily in order to assess their compliance with study intervention. Subjects who are compliant during the single-blind placebo run-in period (subjects must have ≥80% compliance by pill count) will be randomly assigned in a 1:1 ratio to canagliflozin or matching placebo group and will enter the double-blind treatment phase at the randomization visit (Day 1). Subjects randomized to canagliflozin will receive 100 mg canagliflozin, to be taken once daily (QD). After randomization, subjects will return to the clinic at Week 3, Week 13, Week 26, and every 26 weeks thereafter for laboratory assessments, concomitant medication review, adverse event collection and determination of clinical endpoints. At Week 39 and at the midpoint between office visits after Week 52, telephone contact will be made to check the subject status, including discussing study diary entries (ie, collection of self-monitoring of blood glucose (SMBG) and possible hypoglycemic event information), concomitant medication use, adverse events, and determining clinical endpoints (ie, all local laboratory data related to serum creatinine and eGFR). All subjects treated

by the investigator will be managed to reach their glycemic, blood pressure and lipid goals according to established local and regional guidelines, with medical therapies used according to approved local labels. A post-treatment follow-up contact will take place following the treatment phase. Subjects who discontinue study medication prematurely should continue to attend all subsequent study visits and be followed to the global trial end date (GTED). This event-driven study is estimated to have a total duration of approximately 5 to 5.5 years.

A Diagram of the study design is provided below:

Figure 1:



ACEi = angiotensin-converting enzyme inhibitor; UACR = urinary albumin-to-creatinine ratio; AHA = antihyperglycemic agent; ARB = angiotensin receptor blocker; BP = blood pressure; eGFR = estimated glomerular filtration rate;  $HbA_{1c}$  = hemoglobin  $A_{1c}$ ; R = randomization; T2DM= type 2 diabetes mellitus; Wk=week.

# 1.3. Statistical Hypothesis for Trial Objectives

Canagliflozin reduces the risk of the composite endpoint of ESKD, doubling of serum creatinine, and renal or CV death, relative to placebo, in subjects with T2DM, Stage 2 or 3 CKD and

macroalbuminuria, who are receiving standard of care including a maximum tolerated labeled daily dose of an ACEi or ARB.

## 1.4. Sample Size Justification

This is an event driven study. A total of approximately 4,200 subjects will be randomized to either canagliflozin 100 mg or matching placebo in a 1:1 ratio. The study aims to observe the occurrence of the primary efficacy events in 844 unique randomized subjects, on or before the GTED, to have 90% power to detect a 20% relative risk reduction (RRR, defined as one minus hazard ratio) accounting for the effect of treatment discontinuation on the primary endpoint at a 5%, 2-sided significance level.

The above sample size is estimated based on the following additional assumptions:

- Event rate for the composite endpoint in the placebo arm: 6.5% per year
- Premature discontinuation rate of study drug: 6% per year
- Overall lost-to-follow-up: 1%
- Duration of enrollment period: 27 months
- Duration of study (from first subject randomized to last end of study visit): estimated to be 60 months

This is an event driven trial and in order to ensure the number of events are obtained, the study duration and follow-up may be modified, if necessary, based on the observed event rate.

### 1.5. Randomization, Blinding, and Stratification

Upon successful completion of screening, eligible subjects will enter a 2-week run-in period, during which they will receive single-blind placebo capsules (one capsule to be taken once daily before the first meal of the day) to assess compliance with study intervention.

Subjects who are compliant during the single-blind placebo run-in period will be randomly assigned in a 1:1 ratio to canagliflozin 100 mg or matching placebo to be taken once daily, before the first meal of the day. All study intervention after randomization will be provided in a double-blind manner.

Eligible subjects will be stratified according to their screening eGFR ( $\geq$ 30 to <45,  $\geq$ 45 to <60,  $\geq$ 60 to <90 mL/min/1.73m<sup>2</sup>), and will be randomized within the strata.

#### 2. GENERAL ANALYSIS DEFINITIONS

# 2.1. Analysis Populations

- Randomized subjects—subjects who are randomized via the Interactive Web Response System (IWRS);
- Treated subjects—randomized subjects who receive at least one dose of double-blind study medication.

For efficacy analyses and baseline summaries, subjects will be analyzed according to their randomization assignment. For safety analysis (eg, adverse events [AEs]) and summary of exposure, subjects will be analyzed according to the predominant treatment received (defined as the treatment to which the subject was exposed for the greatest duration), in the event that subjects receive a treatment other than the one to which they were randomized. The treatment groups in this SAP will be referred to as canagliflozin and placebo.

# 2.2. Analysis Sets

Analysis sets consist of 2 components: 1) analysis population (Section 2.1), which specifies the subjects included in an analysis; 2) data period, defining the time window during which data will be included in the analysis.

**Table 1:** Summary of Analysis Sets

| Analysis Set | Analysis Population | Data Period |
|---|---|---|
| ITT | Randomized subjects | Day 1 to the last trial contact date (see Section 2.3.1) up to the GTED <sup>a</sup> |
| On-Study | Treated subjects | Day 1 to the last trial contact date (see Section 2.3.1) up to GTED <sup>a</sup> |
| On-Treatment | Treated subjects | Day 1 to the last dose date (see Section 2.3.1) plus X <sup>b</sup> days or the last trial contact date, whichever is earlier. |

For each subject, data collected up to the final visit will be used for analysis. If the final visit can't be arranged, the reported data such as public search of mortality will be bounded by the GTED.

#### 2.3. Time-to-Event Data

### 2.3.1. Subject-Level Trial Milestone Dates

Trial reference start date (Day 1): the first dose date for each subject.

First dose date: the date on which the first dose of study intervention is taken by the subject. If missing or incomplete, the first dose date will be imputed as the randomization date.

Last dose date: the date on which the last dose of study intervention is taken by the subject. If only the day is missing, impute the last day of the month. If the month or the year is missing,

<sup>&</sup>lt;sup>b</sup> X is 2 days for laboratory and vital sign measurements, and 30 days for adverse events (AEs), CV, renal, and mortality endpoints.

impute the date as the date of the scheduled visit after the last visit when the study intervention was dispensed. The imputed last dose date should be no later than the end of treatment visit date or the last trial contact date. In addition, imputed last dose date should be no earlier than the first dose date. The last dose date is the date of permanent study intervention discontinuation regardless of any temporary drug interruption.

Last trial contact date: the date when the last trial-related procedure is conducted. It is defined as the latest of:

- The date of last visit (scheduled or unscheduled visit; office or phone visit), or
- The latest known date of an adverse event (AE) or the study endpoint event status, concomitant medication (CM), vital sign measures (VS) or lab results (LB) as reported on their respective electronic case report from (eCRF) page, or
- The date of alternate contact made (eg, family members, relatives, friends, health care providers) confirming patient was alive at the time of GTED announcement.

For subjects who die during the study or are lost to follow-up, or withdraw consent before announcement of GTED, the last trial contact date will be defined as the date of death or lost to follow-up, or withdrawal of consent. In addition, for subjects who are lost to follow-up, or withdraw consent, where permissible, the available subsequent survival information from a locator agent or public record search will be used to determine the last contact date.

Serum Creatinine Event dates: A doubling of serum creatinine event is defined to occur when a serum creatinine measurement obtained at a post-baseline protocol visit is greater than or equal to twice the baseline average serum creatinine (ie, average value derived from the Day 1 value and the value immediately preceding the Day 1 determination, if both values are available; in addition, the screening value will be used as baseline if all other pre-treatment values are missing). Doubling is confirmed by repeat central laboratory measure after 30 days and preferably within 60 days after the index event and adjudicated as an endpoint event by a blinded Independent Endpoint Adjudication Committee (IEAC). Similarly, an endpoint of ESKD is defined to occur when an eGFR is < 15 ml/min/1.73m<sup>2</sup> based on a serum creatinine obtained at a post-baseline protocol visit, confirmed by repeat central laboratory measure after 30 days and preferably within 60 days after the index event and adjudicated as an endpoint event by the IEAC. In both cases, the date of the event will be defined as the date of the blood draw for the initial serum creatinine measurement (either by local or central laboratory) triggering the event and subsequent adjudication (see Section 5.1.2). If the confirmatory value for doubling of serum creatinine or eGFR < 15 ml/min/1.73m<sup>2</sup> is not available, the endpoint confirmation will be based on the IEAC determination of the event.

## 2.3.2. Censoring Rules

For each analysis set, events that occur any time during the data period of the corresponding analysis set (see Table 1) will be considered as eligible events; otherwise subjects not experiencing an event will be censored at the earlier of their last trial contact day or end of the respective data period, if not otherwise specified.

#### 2.4. Visit Windows

The Time and Events Schedule of the protocol indicates the visit timing and procedures (eg, laboratory, vital signs, and other key safety variables) for each visit; however, the timing of a subject's actual visit may not be exactly as per the protocol indicated target day / visit window. Consequently, for by-visit or over-time summaries, depending on the time period(s) involved in the summaries, the conventions outlined below will be used to allocate the data collected at each actual visit to a planned protocol visit by defining visit windows.

The reference start day is study Day 1 which is the first dose day for subjects who took at least one dose of study medication or the randomization day for subjects who were randomized but did not take any study medication.

Baseline will be defined as the pre-dosing measurement closest to or including Day 1 (prior to dose administration). If the pre-dosing measure on Day 1 is missing, the missing value will be imputed by the latest available measurement prior to Day 1. For serum creatinine, the average of the last two pre-dose measurements will be used as baseline.

If a subject has 2 or more actual visits in one analysis visit window, the visit closest to the target day will be used as the study visit for that analysis visit window. However, results from all visits will be included in the safety analyses (eg, pre-defined limits of change analysis) to ensure that all on-treatment results are included. If 2 study visits are the same number of days from the target day within the same visit window, the later visit will be considered the study visit for that target day. Even though all visits will be allocated an analysis visit window, only planned protocol visits for each variable will be presented in the by-visit analyses.

Note the algorithms for calculating visit windows are the same for all the data periods (see Table 1). Table 2 summarizes the analysis visit windows for laboratory, vital signs, physical examination, and other key safety variables.

**Table 2: Time Intervals for Analysis Visit Windows** 

| Scheduled In-Clinic Visit Time | Time Interval (Day) <sup>a</sup> | Target Time Point (Day) <sup>a</sup> |
|---|---|---|
| Baseline | ≤1 <sup>b</sup> | 1 |
| Week 3 | 1°-56 | 22 |
| Week 13 | 57-137 | 92 |
| Week 26 | 138-229 | 183 |

| Week 39 | 230-320 | 274 |
|------------|-----------|------|
| Week 52 | 321-456 | 365 |
| Week 78 | 457-638 | 547 |
| Week 104 | 639-821 | 730 |
| Week 130 | 822-1003 | 912 |
| Week 156 | 1004-1186 | 1095 |
| Week 182 | 1187-1368 | 1277 |
| Week 208 | 1369-1551 | 1460 |
| Week 234 | 1552-1733 | 1642 |
| Week 260 | 1734-1916 | 1825 |
| Week 286 | 1917-2098 | 2007 |
| Week 312 d | 2099-2281 | 2190 |
| Week 338 d | ≥2282 | 2373 |

- <sup>a</sup> Relative to the day of the first dose of double-blind medication.
- b Up to the first dose of double-blind medication.
- Immediately following the first dose of double-blind medication. For variables without time or reference collected at baseline, the first window after baseline starts on Day 2 according to the protocol.
- d In case the duration of the study goes longer based on the observed event rate.

### 3. INTERIM ANALYSIS

An interim analysis will be conducted when the mean duration of follow-up is at least 2 years and primary efficacy events have been adjudicated as endpoints in approximately 405 subjects. An Independent Data Monitoring Committee (IDMC) will review results of the planned interim analysis and make a recommendation whether the study should be continued as planned, modified, or terminated prematurely due to efficacy, futility or safety reasons.

The analysis method for the primary efficacy endpoint described in Section 5.2 will be used for the interim analysis. The alpha spent in the interim analysis for the testing of the primary composite endpoint is 0.01 (two-sided) which is determined by the alpha spending function taking the form of  $\alpha \tau^{\phi}$  with  $\tau$  as the information fraction and  $\phi = 2.19$ .

The decision rules that trigger the IDMC to consider the recommendation of early study termination will be based on assessment of the primary composite endpoint as well as a "hard" composite endpoint of end-stage kidney disease (ESKD), renal death, and CV death, as specified below:

- Stop the study for efficacy, if the p-value (two-sided) of the primary composite endpoint comparison is <0.01, and the p-value (two-sided) of the composite endpoint of ESKD, renal death, and CV death comparison is <0.025 in favor of canagliflozin. (Note: both composite endpoints must meet their respective efficacy standards for the study to be prematurely terminated for efficacy)
- Stop the study for futility, if the conditional power (based on the assumption that the hazard ratio in the remaining study is 0.80) for achieving the primary composite endpoint at the completion of study is <10% and that the overall benefit profile taking into account both efficacy and safety would be unlikely to be positive at the final analysis of study completion.
- Otherwise continue the study.

If the IDMC recommends early study termination due to efficacy, the sponsor will consider announcing the global trial end date (GTED) and final clinical visits will be scheduled. The test of the primary and the secondary endpoints will be based on the data accrued through the last trial contact date up to the GTED (see Table 1).

#### 4. SUBJECT INFORMATION

### 4.1. Baseline Anthropometric and Demographic Characteristics

Baseline anthropometric and demographic characteristics will be summarized by treatment group and overall (both treatments pooled together) for the ITT analysis sets. Descriptive statistics (N, mean, SD, median, and range) will be provided by treatment group and overall for continuous variables such as age, body weight, and BMI at baseline.

The number and percentage of subjects in the categories of the following variables at baseline will also be summarized by randomized treatment group:

- Age group: <55, 55 to <65, 65 to <75,  $\ge 75$  years old
- Sex: Male, Female
- Race: White, Black or African American, Asian, Others
- Ethnicity: Hispanic or Latino, Not Hispanic or Latino, Unknown, Not reported
- Baseline BMI category: <30, and  $\ge 30 \text{ kg/m}^2$
- Region: North America, Central/South America, Europe, Rest of the World [ROW].

#### 4.1.1. Baseline Disease Characteristics

Descriptive statistics (N, mean, SD, median, and range) will be provided by treatment group and overall for the ITT analysis sets including baseline HbA<sub>1c</sub>, duration of diabetes (in years), baseline eGFR, baseline UACR, baseline SBP/DBP, and baseline status of nicotine use.

The number and percentage of subjects will be summarized by treatment group and overall for the following:

- Baseline HbA<sub>1c</sub> categories: <7%,  $\ge 7\%$  to <8%,  $\ge 8\%$
- Baseline eGFR categories:  $<45, \ge 45$  to  $<60, \ge 60$  mL/min/1.73m<sup>2</sup>
- Baseline UACR categories: ≤1000, >1000 mg/g

The number and percentage of subjects with the complications of diabetes (any and by specific complication) at baseline will be summarized by treatment group and overall. The categories of the complications of diabetes include diabetic retinopathy, autonomic neuropathy, peripheral diabetic neuropathy, other diabetic neuropathy.

In addition to providing results by specific complication, the number and percentage of subjects with at least 2 diabetic complications and all 3 diabetic complications (retinopathy, neuropathy, or nephropathy) will be summarized by treatment group and overall.

The number and percentage of subjects with history of medical conditions by system organ class and preferred term (based upon the general MH eCRF) will be summarized by treatment group and overall. In addition, the following pre-treatment conditions will also be summarized by treatment group and overall.

- Cardiovascular disorders
- Fractures
- Surgeries/Procedures

## 4.2. Disposition Information

Subject disposition will be summarized by treatment group and overall using the following:

- Screen failure
- Subjects who are randomized (ITT analysis set)
- Subjects who are treated
- Subjects who prematurely discontinued study medication prior to the announcement of the GTED

- Subjects who completed the study (ie, defined as having been followed until a time point between the announcement of the GTED and the GTED, or if the subject had died prior to the GTED)
- Subjects without final vital status

Incidences of premature discontinuation from the double-blinded study intervention and the proportion of time on treatment relative to the follow-up period will be provided by treatment group. Time to premature discontinuation from the double-blinded study intervention will be summarized by treatment group using the Kaplan-Meier method.

Listings will be provided for subjects whose predominant treatment differs from their randomized treatment and for subjects who temporarily took the wrong study medication.

# 4.3. Extent of Exposure and Follow-Up

Treatment duration is defined as the amount of elapsed time between the first and the last day that study medication was taken (inclusive). It will be calculated (in days) in terms of the difference in relative study days between the last and first dose of study medication, plus one day.

Follow-up time is defined as the number of days from Day 1 to the last trial contact day (inclusive) for each subject.

Descriptive statistics (N, mean, standard deviation, median, and range) will be presented by treatment group for treatment duration and follow-up.

#### 4.4. Prior and Concomitant Medications

Prestudy (ie, medications taken before initiation of double-blind study medication) and concomitant medications (ie, medications taken after initiation of double-blind study medication that were either started prior or after initiation of double-blind study medication) including AHAs, ACE inhibitors and ARBs, and all other medications are collected.

All prestudy and concomitant medications are coded using World Health Organization Drug Utilization Research Group (WHODRUG) and Anatomical Therapeutic Chemical (ATC) codes.

Prestudy and concomitant medications will be summarized by the number of subjects taking pre-specified categories of medications by treatment group and overall.

The proportion of subjects on ARBs and ACEs, anti-thrombotics (including aspirin) and statins (ie, HMG-CoA reductase inhibitors) at baseline will be summarized by treatment groups based on pre-specified categories (Attachment 1). The proportion of subjects on a maximum labeled dose of ARBs and ACEs for diabetic nephropathy or hypertension at baseline, and the reasons for subjects not on a maximum labeled dose will be summarized. In addition, non-study drug SGLT2 inhibitor use during the follow-up period will be summarized by treatment group.

### 4.5. Patient Management of Cardiovascular Risk Factors

The proportion of subjects with  $HbA_{1c}$  <7% and < 8%, SBP < 140 mm Hg, LDL-C < 100 mg/dL, and the proportion of subjects on statins and on anti-thrombotics (including aspirin) will be summarized by treatment group at Week 52, Week 104, Week 156, Week 208 and Week 260. In addition, longitudinal plots of the mean changes from baseline to the end of study in  $HbA_{1c}$  and SBP will be presented.

### 5. EFFICACY

The primary analysis and major secondary analyses will be performed based on the ITT analysis set.

# 5.1.1. Level of Significance

Unless otherwise specified, all statistical tests except those for the primary efficacy endpoint and major secondary efficacy endpoints, will be interpreted at a 2-sided significance level of 5% and all confidence intervals at a 2-sided confidence level of 95%.

At the interim analysis, the primary efficacy endpoint will be tested with alpha of 0.01 as determined by the alpha spending function taking form of  $\alpha \tau^{\phi}$  with  $\tau$  as the information fraction and  $\phi = 2.19$ .

If the IDMC recommends early study termination due to efficacy, the sponsor will consider announcing the global trial end date (GTED) and final clinical visits will be scheduled. The test of the primary composite endpoint will be based on the data accrued through the final clinic visit where the significance level will be determined by the alpha spending function (Lan et al, 2003 [1]).

If the IDMC does not recommend early study termination, the study will be continued until the target of 844 events have accrued. The primary composite endpoint will be tested with alpha of 0.045 in the final analysis.

Testing of the secondary efficacy endpoints will be based on the data accrued through the final clinic visit (regardless if the study stops after the interim analysis or proceeds to the planned completion of 844 primary composite events) using a two-sided alpha of 0.038. The overall type I error rate will be controlled at the 5% level across the primary and major secondary endpoints using a closed testing procedure, which is detailed in Section 5.5.

# 5.1.2. Data Handling Rules

Unless otherwise stated, all efficacy analyses will be based on the events and the dates identified by the IEAC. The onset of events of doubling of serum creatinine will be confirmed by a central laboratory value after 30 days and preferably within 60 days after the initial doubling. The date of the first documented doubling of serum creatinine will be considered as the onset date of the

event, with the confirmatory value reported by the central laboratory captured as serum creatinine value for the event.

## 5.2. Primary Efficacy Endpoint

### 5.2.1. Definition

The primary efficacy endpoint is the composite endpoint of ESKD, doubling of serum creatinine, and renal or CV death.

Definitions for each component of the primary composite endpoint are:

- ESKD: Initiation of maintenance dialysis for at least 30 days, or renal transplantation, or a eGFR of <15 mL/min/1.73m<sup>2</sup> (by CKD-EPI formula; sustained and confirmed by repeat central laboratory measure after at least 30 days and preferable within 60 days)
- Doubling of serum creatinine: from the baseline determination (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferable within 60 days)
- Renal death: death in patients who have reached ESKD, die without initiating renal replacement therapy, and no other cause of death is determined via adjudication.
- CV death: includes death due to MI, stroke, heart failure, sudden cardiac death, death during
  a CV procedure or as a result of procedure-related complications, or death due to other CV
  causes. For analytic purposes, undetermined causes of death will be considered CV deaths.
  In determining whether a death event is CV in nature, the endpoint adjudication committee
  will take into consideration both the proximate and underlying causes.

For subjects who have ESKD and doubling of serum creatinine determined to have occurred on the same date by the IEAC, the ESKD will be counted as the component for the primary composite endpoint.

### 5.2.2. Analysis Methods

Based on the time from study Day 1 to the first occurrence of the primary efficacy endpoint, the objective of the primary efficacy analysis is to establish that canagliflozin is superior to placebo, in the reduction of the rate of occurrence of the primary efficacy composite endpoint, in subjects with T2DM, Stage 2 or 3 CKD and macroalbuminuria, who are receiving standard of care including a maximum tolerated labeled daily dose of an ACEi or ARB.

The hypothesis of the superiority on the primary efficacy endpoint for the comparison of canagliflozin versus placebo will be analyzed using a stratified Cox proportional hazard model including treatment, with stratification of the baseline hazard by screening eGFR (<45,  $\ge45$  to <60,  $\ge60$  mL/min/1.73m<sup>2</sup>). The primary analysis will be based on the ITT analysis set from study

Day 1 up to the GTED. If the study is not stopped prematurely for efficacy based on the interim analysis, the superiority will be evaluated at the final analysis using a 2-sided test with  $\alpha$ =0.045.

Estimates of the RRR (defined as one minus the hazard ratio), the hazard ratio and corresponding 95% CIs will be provided.

## 5.2.2.1. Supportive Efficacy Analyses

The cumulative incidence of the primary efficacy composite over time will be presented using Kaplan-Meier curves for each of the 2 treatment groups. Cumulative incidence curves will also be presented for each of the components of the primary composite (ESKD, doubling of serum creatinine, renal death, and CV death) in order to assess competing risks, depending on the event counts of the individual components.

In addition, ratios of cause-specific hazards between the treatment groups will be obtained for each component of the primary efficacy composite endpoint (ESKD, doubling of serum creatinine, renal death, or CV death), with stratification of the baseline hazard by screening eGFR group as in the analysis of the primary efficacy composite.

To assess the robustness of the primary efficacy analysis, sensitivity analysis of the primary efficacy endpoint using a log-rank test stratified by screening eGFR will also be performed. The log-rank test does not require the proportional hazards assumption as for Cox proportional hazard model.

Extensive efforts will be made to collect complete event and vital status data for all subjects randomized in this study. To illustrate the extent of missingness for the primary efficacy endpoint, the numbers of subjects with missing follow-up and the percentages of total missing follow-up time vs total number of subjects randomized and expected follow-up time will be summarized. Missing follow-up time for subjects who did not die will be calculated from last contact date to the announcement of GTED. For each subject, expected follow-up time will be calculated from study Day 1 to the earliest date of announcement of GTED or first occurrence of the primary efficacy endpoint.

An On-Treatment analysis (which includes composite endpoints with an onset after the initiation of double-blind study medication and before the last study medication date + 30 days) will also be performed to assess the consistency of the primary efficacy analysis. This will use a similar analysis model to the primary analysis.

# 5.2.2.1. Assessment of Model Assumption in the Primary Efficacy Analysis

The proportional hazards assumption for the primary efficacy analysis model will be assessed graphically using Log (-log) plots and/or plots of Schoenfeld residuals. In addition, a linear non-proportionality test will be performed. If evidence of deviations from the proportional hazards assumption is detected, additional Cox regression analyses with time-dependent hazard

ratios for the treatment effect may be explored to better understand the degree and nature of the treatment effect differences over time.

## 5.3. Subgroup Analyses for the Primary Endpoint

The homogeneity of treatment effects on the occurrence of the primary efficacy endpoint across subgroups (if a total number of events is greater than 10 for both treatment groups and at least 1 event in both groups) will be examined (at a 2-sided significance level of 0.10) via a test for the treatment by subgroup interaction by adding this term and the subgroup as covariates (viewed as class variables) to the primary efficacy analysis model. Factors exhibiting interactions with p < 0.10 will be identified as exhibiting a possible treatment effect heterogeneity, recognizing that one or more p-values under 0.10 may be expected to be observed by chance when multiple subgroup factors are examined.

If a significant interaction is observed, the results will be examined to determine whether the interaction is qualitative. If the interaction is qualitative in nature, clinical explanations of the significant interaction will be explored.

Estimates and 2-sided 95% confidence intervals for the hazard ratio (canagliflozin/placebo) will be provided for each subgroup. The analyses will be based on the primary efficacy analysis model separated for each subgroup.

The subgroups are listed below:

- Sex: male or female
- Age group: <65, ≥65 years old</li>
- Race group: White, Black or African American, Asian, Other
- Ethnicity: Hispanic or Latino, Not Hispanic or Latino, Not reported/Unknown
- Region: North America, Central/South America, Europe, and ROW
- Duration of diabetes at baseline <median or ≥ median years
- CV history at baseline: Yes, No
- Baseline BMI:  $<30 \text{ or } \ge 30 \text{ kg/m}^2$
- Baseline HbA<sub>1c</sub> categories: <8%, ≥8%
- Baseline eGFR:  $<45, \ge 45$  to  $<60, \ge 60$  mL/min/1.73m<sup>2</sup>
- Baseline UACR categories: ≤1000, >1000 mg/g
- Baseline SBP categories: ≤ the median, > the median

• History of amputation: Yes, No

# 5.4. Major Secondary Endpoints

### 5.4.1. Definition

Major secondary efficacy endpoints include:

- Composite endpoint of CV death and hospitalized congestive heart failure
- Composite endpoint of CV death, non-fatal MI, and non-fatal stroke (ie, 3-point MACE)
- Hospitalized congestive heart failure
- Renal composite endpoint of ESKD, doubling of serum creatinine, and renal death
- CV death
- All-cause death
- CV composite endpoint of CV death, non-fatal MI, non-fatal stroke, hospitalized congestive heart failure, and hospitalized unstable angina

# 5.4.2. Analysis Methods

If superiority of canagliflozin over placebo in reducing the risk of the primary efficacy endpoint is established, the hypothesis of superiority on major secondary efficacy endpoints of canagliflozin versus placebo will be subsequently tested in the following hierarchical order:

- 1. Composite endpoint of CV death and hospitalized congestive heart failure
- 2. Composite endpoint of CV death, non-fatal MI, and non-fatal stroke (ie, 3-point MACE)
- 3. Hospitalized congestive heart failure
- 4. Renal composite endpoint of ESKD, doubling of serum creatinine, and renal death
- 5. CV death
- 6. All-cause death
- 7. CV composite endpoint of CV death, non-fatal MI, non-fatal stroke, hospitalized congestive heart failure, and hospitalized unstable angina

Time from study Day 1 to the first occurrence of a major secondary efficacy endpoint will be analyzed using the same approach as the primary analysis based on the data scope from study Day 1 to GTED in the ITT analysis set.

# 5.5. Multiplicity Adjustment

A closed testing procedure will be implemented to control the family-wise type I error rate at 5% for primary and secondary endpoints. The hypothesis of superiority on primary and major secondary efficacy endpoints of canagliflozin versus placebo will be tested in the following hierarchical order. If an individual test during any step is not statistically significant, later tests will not be declared to be statistically significant.

Figure 2: Hypothesis Testing Sequence



<sup>\*</sup> If IDMC recommends early study termination due to efficacy, the primary composite endpoint will be tested after final study visit for the last subject completed the study, with the significance level determined by the accrued events and the alpha spending function.

# 5.6. Other Efficacy Analyses

### 5.6.1. Definition of Exploratory Efficacy Endpoints

In addition to the primary and major secondary endpoints previously described, the following endpoints and measurements will also be analyzed:

- 1. Composite endpoint events of ESKD (defined as a sustained eGFR of <15 mL/min/1.73m<sup>2</sup> or initiation of dialysis with maintenance for at least 30 days, or renal transplantation) and CV death or renal death
- 2. Individual components of the renal and cardiovascular composite endpoints (ESKD, doubling of serum creatinine, renal death, CV death, fatal or non-fatal MI, fatal or non-fatal stroke, hospitalized congestive heart failure, hospitalized unstable angina)
- 3. Changes in estimated glomerular filtration rate (eGFR) over time
- 4. Changes in urinary albumin-to-creatinine ratio (UACR) over time

# 5.6.2. Definition of Other Efficacy Endpoints

- 1. Composite endpoint events of ESKD (defined as a sustained eGFR of <15 mL/min/1.73m<sup>2</sup> or initiation of dialysis with maintenance for at least 30 days, or renal transplantation) and renal death
- 2. Composite endpoint events of ESKD (defined as a sustained eGFR <15 mL/min/1.73m<sup>2</sup> with symptoms of uremia or a sustained eGFR of <8 mL/min/1.73m<sup>2</sup> or initiation of dialysis with maintenance for at least 30 days, or renal transplantation) and CV death or renal death
- 3. Composite endpoint events of ESKD (defined as a sustained eGFR <15 mL/min/1.73m<sup>2</sup> with symptoms of uremia or a sustained eGFR of <8 mL/min/1.73m<sup>2</sup> or initiation of dialysis with maintenance for at least 30 days, or renal transplantation) and renal death

## 5.6.3. Analysis Methods for Other Efficacy Analyses

### Composite endpoint events (described in Section 5.6.1)

The time from study Day 1 to the first occurrence of composite endpoint events in each of the aforementioned composites will be analyzed by a method similar to that used for the primary efficacy analysis based on the data scope from study Day 1 to GTED in the ITT analysis set.

### eGFR change over time

The on-treatment eGFRs include all central laboratory eGFR measurements from study Day 1 up to the last dose plus 2 days. The change from baseline in eGFR will be analyzed using a restricted maximum likelihood (REML) repeated measures approach. The analysis will be based on observed data and will include the fixed, categorical effects of treatment, stratification factor, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline eGFR and baseline-by-visit interaction. An unstructured covariance will be used to model the within-patient errors. The adjusted mean changes in eGFR from baseline will be plotted over time by treatment group to depict the pattern of change in mean eGFR over time. Linear contrasts will be constructed to estimate the treatment effect on the mean change in eGFR to

6 months (early effect), the mean change in eGFR from 6 months to 4 years (late effect), and the mean change in eGFR from baseline to 4 years (overall effect).

If the changes in mean eGFR in the above analysis exhibit a linear trajectory after 6 months, a multi-slope mixed effects linear spline model will be fitted with separate slopes from baseline to month 3, from month 3 to month 6, and from month 6 to the GTED. This model will be constructed with fixed effects for the screening eGFR randomization strata and with random intercepts and slopes to account for variation in progression rates over time. Likelihood based comparisons of goodness of fit will be used to determine if the model should be expanded to include additional terms to account for auto-correlation in residual over time, differences in variance between the treatment and control groups, or other deviations from the random slope-intercept model. The mean slopes from baseline to month 3 and from baseline to month 6 will be compared between the treatment groups to estimate the immediate and longer term acute effects of canagliflozin vs. placebo. The long-term slopes after month 6 will be used to estimate the effect of canagliflozin on the "chronic" slope after 6 months. The estimated mean change in eGFR from baseline to 4 years will also be compared under the 3 slope model to estimate the overall effect of canagliflozin on the mean change in eGFR.

A similar analysis based on all central laboratory eGFR measurements from study Day 1 up to the end of study will be conducted using the similar model.

If the distribution of eGFR value is positively skewed, log transformation of eGFR values may be considered prior to the modeling.

### **UACR** change over time

On-treatment central laboratory UACR will be analyzed using the similar model for eGFR. Log transformation of UACR values will be made prior to the modeling, since the distribution of UACR value is highly skewed.

A similar analysis for UACR measurements from study Day 1 up to the end of study will be performed using the similar model.

#### 6. SAFETY

Treatment-emergent safety analyses and summaries will be based on the On-Treatment analysis set (Section 2.2). All safety analyses and summaries will utilize this approach unless otherwise specified.

There will be no imputation of missing values for clinical laboratory test results and vital sign measurements in the safety analyses, and there will be no hypothesis testing for results from safety analyses.

The study objective regarding safety and tolerability will be assessed based upon a review of the incidence of all adverse events, as well as laboratory results, and other safety and tolerability measurements.

#### 6.1. Adverse Events

Adverse events (AEs) will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) at the time of database lock. Therefore, the preferred terms presented in Attachment 2 may be modified to reflect such updates. A treatment-emergent AE (TEAE) is defined as an adverse event with an onset after the initiation of double-blind study medication and before the last study medication date + 30 days (ie, the On-Treatment analysis set). AEs with a start date prior to initiation of double-blind study medication which are subsequently reported to have either an increase in intensity or change in attribution in relationship to study medication (ie, no attribution to possible, probably, very likely) after the initiation of double-blind study medication will also be considered as TEAEs.

In addition to treatment-emergent AE analyses for selected AEs with an onset after the initiation of study medication and regardless of time off the study medication will also be performed.

#### 6.1.1. General Adverse Events

An overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- Any AEs
- Serious AEs
- Deaths
- AEs leading to discontinuation of study medication
- Serious AEs leading to discontinuation of study medication
- Serious AEs considered drug-related
- AEs considered drug-related leading to discontinuation of study medication

SAEs and AEs leading to discontinuation of study medication (by system organ class and preferred term) will be summarized by treatment group using the On-Treatment analysis set. AEs by system organ class (ie, number and percent of subjects with one or more AEs within a system organ class) will similarly be summarized by treatment group.

The overall incidence (ie, number and percent of subjects with one or more AE in each category) of AEs, AEs leading to discontinuation, drug-related AEs, drug-related AEs leading to discontinuation of study medication, serious AEs, serious AEs leading to discontinuation, serious drug-related AEs, serious drug-related AEs leading to discontinuation of study medication and deaths, will be summarized by treatment group.

For each AE, the percentage of subjects who experienced at least one occurrence of the given event will be provided by preferred term, grouped by system organ class (SOC), and presented by treatment group. In addition, the incidence of AEs (by preferred term, grouped by SOC, and presented by treatment group) will also be summarized by severity (by each designation, and pooling mild or moderate), by the relationship to study medication, by the action taken regarding the study medication, as well as by the outcome. The relationship to study medication will be presented by 2 categories: related (which includes possibly related, probably related and very likely related, as reported by the investigator) and not related (which includes not related and doubtfully related, as reported by the investigator), as well as by individual designation.

Listings will also be generated for deaths, SAEs, and discontinuations due to AEs.

As a screening tool, the 95% CIs for the percentage difference between canagliflozin and placebo will be provided for the AEs which are reported in at least four or more subjects in any treatment group. Four (rule-of-4) was chosen based on the recommendation from the Safety, Planning, Evaluation, and Reporting Team (SPERT)[2]. No multiplicity adjustment will be applied. The exclusion of "0" in the 95% CI around the difference in incidence for a particular AE does not necessarily imply that the higher incidence is related to drug. The intent of providing the 95% CIs is as a filter to identify AEs that require additional assessment. Adverse events for which there is an imbalance in incidence with 0% in placebo and 0.5% or higher in canagliflozin will be further evaluated.

Adverse events that are identified by the above screening procedure will be subject to further evaluation. The additional assessment may include some or all of the following:

- 1. Investigator assessed relationship of AE to study intervention, investigator assessed intensity of AE
- 2. Time to AE relative to start of double-blind study medication, duration of AE, action taken on study intervention/occurrence of AEs leading to discontinuation
- 3. Other relevant safety information such as observations in other canagliflozin trials, observations in trials of other members of the SGLT2 inhibitor class, biological plausibility of the AE as related to SGLT2 inhibition or to canagliflozin.

#### 6.2. Adverse Events of Interest

In order to support the additional assessment of particular categories of adverse events, such as fractures and volume depletion, medical queries of selected preferred terms have been created. A blinded review prior to database lock will be performed to ensure that no reported term suggestive of the AE of interest is omitted. The list of preferred terms that are to be combined for the assessment of each of the pre-specified adverse events (eg, malignancies, severe hypersensitivity reactions [eg, angioedema, anaphylaxis, Stevens-Johnson syndrome], photosensitivity reactions, serious adverse events of hepatic injury, nephrotoxicity/acute kidney

injury, venous thromboembolic events, diabetic ketoacidosis [DKA], pancreatitis, fractures, and amputation) are provided in Attachment 2. The primary analysis of DKA, pancreatitis, and fracture will be based on adjudication results. Selected adverse events (eg, DKA, amputation, malignancy, and fracture) will be performed in both On-Treatment and On-Study analysis sets.

The incidences and descriptive statistics of the additional information collected for each AE of interest will be summarized by treatment group. Additionally, the percentage of subjects with each AE of interest will be summarized by severity and relationship to study intervention. Treatment differences in incidence rates and corresponding 95% CI will be provided.

The Kaplan-Meier plots for the time to first occurrence by treatment group will also be generated for certain AEs such as adjudicated fractures and amputation AEs. The time to first occurrence of the AE will be defined as the number of days between the study Day 1 and the onset day of the first occurrence. Subjects without the AE will be censored at the last dose date plus 30 days or the last trial contact date as defined in Section 2.2, whichever is earlier.

#### 6.3. Modified Rankin Scores for Stroke

The ordinal categories of modified Rankin scores for the events of stroke will be summarized by treatment group based on investigator's assessment. The modified Rankin score will be grouped to the ordered categories: 0-2 = nondisabling, 3-5 =disabling, 6 =death. For adjudicated stroke cases, the change of the score before and after the event will be calculated and used to assess the severity of the event.

# 6.4. Hypoglycemia

All hypoglycemic episodes are to be reported on an eCRF page specific for hypoglycemia. If the hypoglycemia episode is considered to be an AE/SAE in the opinion of the investigator, the episode is also to be recorded on the AE/SAE eCRF page. Hypoglycemia as AEs/SAEs will be presented in the tabulation of AEs described above. All additional analyses of hypoglycemia episodes will be based on results collected using the hypoglycemia eCRF. Reconciliation will be conducted to ensure that all hypoglycemia episodes reported as AEs are also recorded on the hypoglycemia eCRF form; however, hypoglycemia episodes reported on the hypoglycemia eCRF do not have to be reported as an AE (deferred to the investigator's determination). Analyses discussed below are based upon episodes reported through the hypoglycemia eCRF.

A subject will be counted as having a documented hypoglycemia episode when there is either a biochemically confirmed hypoglycemic episode (ie, concurrent fingerstick glucose or plasma glucose ≤70 mg/dL (3.9 mmol/L), and/or a severe hypoglycemic episode, as reported on the hypoglycemia eCRF, as follows:

• Biochemically documented hypoglycemia episode: a hypoglycemia episode with a concurrent reported glucose value of ≤70 mg/dL (3.9 mmol/L), regardless of whether the

episode is associated with symptoms (symptomatic hypoglycemia) or not (asymptomatic hypoglycemia)

• Severe hypoglycemia episode: a hypoglycemia episode that has the answer "Yes" recorded for any of the following 3 questions on the hypoglycemia eCRF: "Did the subject require assistance for this episode?", "Did the subject lose consciousness during the episode?", or "Did the subject have a seizure during the episode?"

Only treatment-emergent hypoglycemia episodes (defined the same way as treatment-emergent AEs in Section 6.1) reported on the eCRF for hypoglycemia will be summarized.

The percentage of subjects with documented hypoglycemia episodes (ie, biochemically documented and/or severe) and subjects with biochemically documented, and with severe hypoglycemia episodes separately, will be summarized by treatment group. For subjects with biochemically documented hypoglycemia episodes, the percentage of subjects will be summarized for each of the following glucose levels (≤70 mg/dL [3.9 mmol/L], <56 mg/dL [3.1 mmol/L], and <36 mg/dL [2.0 mmol/L], "Low" results will be included in all three categories) by treatment group. For subjects with severe hypoglycemia episodes, the percentage of subjects by each answer of the 3 questions for severe hypoglycemia on the eCRF will be summarized by treatment group. Event rate by person-year (total number of episodes/total exposure) will be calculated by treatment group separately for documented and for severe hypoglycemia.

Subjects who had 0, 1, 2, or  $\geq 3$  documented episodes and subjects who had 0, 1, 2, or  $\geq 3$  severe hypoglycemic episodes will be summarized by treatment group.

In addition, the incidence of all episodes of hypoglycemia reported on the eCRF for hypoglycemia will be provided (this includes events without concurrent fingerstick glucose reported and events with fingerstick glucose >70 mg/dL [3.9 mmol/L]) by treatment group.

### 6.5. Clinical Laboratory Tests

Laboratory data will be summarized for each type of laboratory test listed in Attachment 3. Normal reference ranges for each test will be provided. Descriptive statistics (N, mean, standard deviation, median, and range, as well as the 95% CI for the change from baseline) will be reported for each laboratory analyte at baseline and at each scheduled time point for absolute value and for change and percent change from baseline. Descriptive statistics will be presented for the On-Treatment analysis set (ie, based on measurements on study medication, including up to a maximum of 2 days after the last dose of study medication) as well as for the On-Study analysis set (ie, all measurements regardless of the time of the last dose of double-blind study intervention). Summaries based on both standard units (SI) and conventional units will be provided.

The percentage of subjects with specific treatment-emergent laboratory values meeting pre-defined limit of change (PDLC) criteria will be summarized for these laboratory analytes. The 95% CI for the percentage difference between canagliflozin and placebo will be provided for each PDLC criterion which have at least 4 or more subjects in any treatment group; a corresponding listing will also be provided. The criteria for PDLC values are listed in Attachment 4.

### 6.6. Vital Signs

Descriptive statistics (N, mean, standard deviation, median, and range, as well as the 95% CI for the change from baseline) will be reported for systolic and diastolic blood pressure (SBP and DBP), and pulse at each scheduled time point for absolute value and for change from baseline. Descriptive statistics will be presented for the On-Treatment analysis set (ie, based on measurements on study medication, including up to a maximum of 2 days after the last dose of study medication) as well as On-Study analysis set (ie, all measurements regardless of the time of the last dose). The blood pressure measurements will be based on the average of the consecutive sitting blood pressure readings that were to be collected at each visit.

A treatment-emergent vital sign abnormality is defined as a change from baseline and subsequent post-baseline value that satisfies the PDLC criteria listed in Attachment 4. For each vital sign parameter, the proportion of subjects with a treatment-emergent abnormality will be tabulated by treatment group. The 95% CI for the percentage difference between canagliflozin and placebo will be provided for each PDLC criterion which have at least 4 or more subjects in any treatment group; a corresponding listing will also be provided.

## **REFERENCES**

- 1. Lan K. K. G., Lachin, J M, and Bautista, O. (2003), Over-ruling a group sequential boundary a stopping rule versus a guideline. Statistics in Medicine 22, 3347–3355.
- Brenda J, Crowe, H etc. Recommendations for safety planning, data collection, evaluation and reporting during drug, biologic and vaccine development: a report of the safety planning, evaluation, and reporting team. Clin Trials 2009 6: 430-440

## **ATTACHMENT 1**

Prestudy and Concomitant Medications Classified by ATC Code and/or Other Conditions

Note: The ATC code might be changed based on the latest version at the time of database lock

| Medication | ATC code and/or Other Conditions |
|---|---|
| Anti-Hyperglycemic<br>Agents (AHA) | ATC Code starts with 'A10' (Drugs used in diabetes) |
| Insulin | ATC Code starts with 'A10A' (Insulins and analogues) |
| Biguanides | ATC Codes start with 'A10BA' (Biguanides); and/or appropriate 'A10BD' (combinations of oral blood glucose lowering drugs) |
| Sulfonamides | ATC Codes start with 'A10BB' (sulfonamides, urea derivatives), 'A10BC' (sulfonamides [heterocyclic]); and/or appropriate 'A10BD' (combinations of oral blood glucose lowering drugs) |
| Alpha glucosidase<br>Inhibitors | ATC Code starts with 'A10BF' (alpha glucosidase inhibitors) |
| Thiazolidinediones (PPARγ) | ATC Codes start with 'A10BG' (Thiazolidinediones); and/or appropriate 'A10BD' (combinations of oral blood glucose lowering drugs) and/or 'A10BX' (other blood glucose lowering drugs, excluding insulins) |
| Dipeptidyl peptidase 4<br>(DDP-4) Inhibitors | ATC Codes start with 'A10BH' (Dipeptidyl peptidase 4 [DPP-4]); and/or appropriate 'A10BD' (combinations of oral blood glucose lowering drugs) |
| GLP 1 | ATC Codes start with 'A10BJ' (other blood glucose lowering drugs, excluding insulins) |
| Glinides | ATC Codes start with appropriate 'A10BD' (combinations of oral blood glucose lowering drugs) and/or 'A10BX' (other blood glucose lowering drugs, excluding insulins) |
| SGLT2i | ATC Code starts with 'A10BK' (with ingredient of 'dapagliflozin', 'canagliflozin', 'empagliflozin', 'dapagliflozin propanediol monohydrate', or 'ertugliflozin') or |
| | ATC Code start with appropriate 'A10BD' (with ingredient of 'canagliflozin, metformin hydrochloride', 'empagliflozin, |

| Medication | ATC code and/or Other Conditions |
|---|---|
| | linagliptin') |
| Other Anti- | ATC Code starts with 'A10BX' (other blood glucose lowering |
| Hyperglycemic Agents | drugs, excluding insulins) |
| Lipid-Altering | ATC Codes start with 'C10' |
| Medications | <ul> <li>Lipid modifying agents, plain</li> </ul> |
| | ATC Codes start with 'C10A' |
| | • Lipid modifying agents, combinations |
| | ATC Codes start with 'C10B' |
| Antihypertensives | Angiotensin-Converting Enzyme Inhibitors (ACEi): ATC Codes start with 'C09A' (ACE inhibitors, plain), and/or 'C09B' (ACE |
| | inhibitors, combinations) with one of the following combination |
| | ingredients containing ACE inhibitors. |
| | Angiotensin-Receptor Blockers (ARB): ATC Codes start with |
| | 'C09C' (Angiotensin II antagonists); and/or 'C09D' (Angiotensin II |
| | antagonists, combinations) with one of the following combination |
| | ingredients containing an angiotensin II antagonist. |

#### 1. DIURETICS

Diuretics (loop) or diuretics (non-loop):

# 1.1. Diuretics [loop]

ATC Codes start with 'C03C' (High-ceiling diuretics), and/or 'C02LA' (Rauwolfia alkaloids and diuretics in combination) with one of the following combination ingredients:

Dihydralazine Sulfate, Furosemide, Reserpine

Dihydralazine Sulfate, Furosemide, Reserpine, Triamterene

Furosemide, Reserpine

and/or 'C03EB' (High-ceiling diuretics and potassium-sparing agents) with one of the following combination ingredients:

Amiloride Hydrochloride, Bumetanide

Amiloride Hydrochloride, Furosemide

Amiloride, Furosemide

Furosemide Xantinol, Triamterene

Furosemide, Spironolactone

Furosemide, Triamterene

Furosemide Sodium, Potassium Canrenoate

and/or 'C09BA' (ACE inhibitors and diuretics) with one of the following combination ingredients:

Furosemide,Ramipril Piretanide,Ramipril

# 1.2. Diuretics [non-loop]

ATC Codes start with 'C03A' (Low-ceiling diuretics, thiazides), 'C03B' (Low-ceiling diuretics, excluding thiazides), 'C03D' (Potassium-sparing agents),

and/or 'C02LA' (Rauwolfia alkaloids and diuretics in combination) with one of the following combination ingredients:

Adonis Vernalis Extract, Benzthiazide, Convallaria Majalis Extract, Drimia Maritima Extract, Oleandrin, Potassium Aspartate, Rauwolfia Serpentina

Ajmaline, Benzylhydrochlorthiazide, Potassium

Chloride, Raupine, Rescinnamine, Reserpine Hydrochloride, Yohimbine

Ajmaline, Benzylhydrochlorthiazide, Potassium

Chloride, Raupine, Rescinnamine, Yohimbine

Ajmaline,Corynanthine,Hydrochlorothiazide,Raupine,Rescinnamine,Rescrpine Hydrochloride

Altizide, Potassium Canrenoate, Rescinnamine

Bemetizide, Potassium Chloride, Pyridoxine

Hydrochloride, Reserpine, Retinol, Thiamine Mononitrate, Tocopheryl Acetate

Bendroflumethiazide, Methiomeprazine, Reserpine

Bendroflumethiazide, Potassium Chloride, Rauwolfia Serpentina

Bendroflumethiazide, Potassium Chloride, Reserpine

Bendroflumethiazide, Rauwolfia Serpentina

Bendroflumethiazide, Reserpine

Benziodarone, Hydroflumethiazide, Potassium Chloride, Reserpine

Benzthiazide, Methoserpidine

Benzthiazide, Reserpine

Benzylhydrochlorthiazide, Carbazochrome, Reserpine

Benzylhydrochlorthiazide, Diisopropylamine Dichloroacetate, Rescinnamine

Butizide, Carbocromen, Potassium Chloride, Raubasine, Rescinnamine, Reserpine

Butizide, Potassium Chloride, Raubasine, Rescinnamine, Reserpine

Butizide, Reserpine, Spironolactone

Chlorothiazide, Dihydralazine Tartrate, Rauwolfia Serpentina

Chlorothiazide, Rescinnamine

Chlorothiazide, Reserpine

Chlortalidone, Dihydralazine Hydrochloride, Oxazepam, Potassium

Gluconate, Protoveratrines A And B, Reserpine, Rutoside, Xantinol Nicotinate

Chlortalidone, Dihydroergocristine, Magnesium Sulfate

Heptahydrate, Methylergometrini Tartras, Reserpine, Thiourea

Chlortalidone, Reserpine

Chlortalidone, Reserpine, Spironolactone

Clofenamide, Reserpine

Clofenamide, Reserpine, Rutoside

Clopamide, Dihydroergocristine Mesilate, Reserpine

Clopamide, Dihydroergocristine, Reserpine

Clopamide, Dihydroergotoxine Mesilate

Clopamide, Reserpine

Cyclopenthiazide, Potassium Chloride, Reserpine

Cyclothiazide, Diprophylline, Methoserpidine

Cyclothiazide, Reserpine

Deserpidine, Hydrochlorothiazide

Deserpidine, Methyclothiazide

Dihydralazine Sulfate, Hydrochlorothiazide, Potassium Chloride, Reserpine

Dihydralazine Sulfate, Hydrochlorothiazide, Reserpine

Dihydralazine, Hydrochlorothiazide, Potassium Chloride, Reserpine

Dihydralazine, Hydrochlorothiazide, Reserpine

Dihydroergotamine Mesilate, Hydrochlorothiazide, Reserpine

Ethiazide, Potassium Chloride, Rauwolfia Serpentina

Flumethiazide, Potassium Chloride, Rauwolfia Serpentina

Guanethidine Sulfate, Hydrochlorothiazide, Methyldopa, Reserpine

Hydralazine Hydrochloride, Hydrochlorothiazide, Reserpine

Hydrochlorothiazide, Mecamylamine Hydrochloride, Neostigmine

Metilsulfate, Rescinnamine

Hydrochlorothiazide, Methoserpidine

Hydrochlorothiazide, Methyldopa, Reserpine, Triamterene

Hydrochlorothiazide, Nicergoline, Reserpine

Hydrochlorothiazide, Pentosan Polysulfate, Rauwolfia Serpentina

Extract, Trichlormethiazide, Xantinol Nicotinate

Hydrochlorothiazide, Potassium Chloride, Rauwolfia

Serpentina, Rescinnamine, Reserpine, Retinol Palmitate, Tocopheryl Acetate

Hydrochlorothiazide, Potassium Chloride, Reserpine

Hydrochlorothiazide, Reserpine

Hydrochlorothiazide, Reserpine, Secbutabarbital

Hydrochlorothiazide, Reserpine, Triamterene

Hydroflumethiazide, Reserpine

Inositol Nicotinate, Mefruside, Rescinnamine

Inositol Nicotinate, Mefruside, Reserpine

Mefruside, Methyldopa, Reserpine

Mefruside, Reserpine

Methyclothiazide, Reserpine

Polythiazide, Reserpine

Quinethazone, Reserpine

Reserpine, Trichlormethiazide

Reserpine, Xipamide

and/or 'C02LB' (Methyldopa and diuretics in combination) with one of the following combination ingredients:

Amiloride Hydrochloride, Hydrochlorothiazide, Methyldopa

Amiloride, Hydrochlorothiazide, Methyldopa

Benzthiazide,Methyldopa Butizide,Methyldopa Chlorothiazide,Methyldopa Hydrochlorothiazide,Methyldopa Mefruside,Methyldopa

and/or 'C02LC' (Imidazoline receptor agonists in combination with diuretics) with one of the following combination ingredients:

Bencyclane Fumarate, Clonidine Hydrochloride, Hydrochlorothiazide

Bendroflumethiazide, Clonidine

Chlortalidone, Clonidine

Chlortalidone, Clonidine Hydrochloride

Chrysanthemum Spp., Clonidine Hydrochloride, Concha

Margaritifera, Hydrochlorothiazide, Rutoside

Clonidine Hydrochloride, Cyclothiazide

Clonidine Hydrochloride, Hydrochlorothiazide, Triamterene

and/or 'C02LF' (Guanidine derivatives and diuretics) with one of the following combination ingredients:

Polythiazide, Prazosin Hydrochloride

Bemetizide, Guabenxan

Cyclopenthiazide, Guanethidine Sulfate

Cyclopenthiazide, Guanethidine Sulfate, Potassium Chloride

Guanethidine Sulfate, Hydrochlorothiazide

Guanoxan Sulfate, Polythiazide

and/or 'C02LG' (Hydrazinophthalazine derivatives and diuretics) with one of the following combination ingredients:

Dihydralazine Tartrate, Hydrochlorothiazide, Mebutamate, Potassium Chloride Hydralazine Hydrochloride, Hydrochlorothiazide

and/or 'C02LK' (Alkaloids, excluding rauwolfia, in combination with diuretics) with one of the following ingredients:

Cryptenamine Tannates, Methyclothiazide

and/or 'C02LL' (MAO inhibitors and diuretics) with one of the following combination ingredients:

Methyclothiazide, Pargyline Hydrochloride

and/or 'C02LX' (Other antihypertensives and diuretics) with one of the following combination ingredients:

Bemetizide, Bupranolol Hydrochloride, Dihydralazine Sulfate, Triamterene

and/or 'C03EA' (Low-ceiling diuretics and potassium-sparing agents) with one of the following combination ingredients:

Altizide, Spironolactone

Amiloride Hydrochloride, Bendroflumethiazide

Amiloride Hydrochloride, Chlortalidone

Amiloride Hydrochloride, Cyclopenthiazide

Amiloride Hydrochloride, Hydrochlorothiazide

Amiloride, Amiloride Hydrochloride, Methyclothiazide

Amiloride, Hydrochlorothiazide

Bemetizide, Hesperidin Complex, Thiamine Mononitrate, Triamterene

Bemetizide, Triamterene

Bendroflumethiazide, Spironolactone

Benzthiazide, Triamterene

Butizide, Potassium Canrenoate

Butizide, Spironolactone

Chlortalidone, Spironolactone

Chlortalidone, Triamterene

Clofenamide, Triamterene

Cyclothiazide, Triamterene

Epitizide, Triamterene

Hydrochlorothiazide, Spironolactone

Hydrochlorothiazide, Triamterene

Hydrochlorothiazide, Triamterene, Verapamil Hydrochloride

Hydroflumethiazide, Spironolactone

Mebutizide, Triamterene

Methyclothiazide, Triamterene

Metolazone, Triamterene

Triamterene, Trichlormethiazide

Triamterene, Xipamide

and/or 'C03EB' (High-ceiling diuretics and potassium-sparing agents) with one of the following combination ingredients:

Amiloride Hydrochloride, Bumetanide

Amiloride Hydrochloride, Furosemide

Amiloride, Furosemide

Furosemide Xantinol, Triamterene

Furosemide, Spironolactone

Furosemide, Triamterene

and/or 'C03XA' (Vasopressin antagonists) with one of the following ingredients or combination ingredients:

Conivaptan

Conivaptan Hydrochloride

Satavaptan

Tolvaptan
and/or 'C09BA' (ACE inhibitors and diuretics) with one of the following combination ingredients:

Benazepril Hydrochloride, Hydrochlorothiazide

Benazepril, Hydrochlorothiazide

Captopril, Hydrochlorothiazide

Cilazapril, Hydrochlorothiazide

Delapril Hydrochloride, Indapamide

Delapril, Indapamide

Enalapril Maleate, Hydrochlorothiazide

Enalapril, Hydrochlorothiazide

Fosinopril Sodium, Hydrochlorothiazide

Fosinopril, Hydrochlorothiazide

Hydrochlorothiazide, Imidapril Hydrochloride

Hydrochlorothiazide, Lisinopril

Hydrochlorothiazide, Lisinopril Dihydrate

Hydrochlorothiazide, Moexipril Hydrochloride

Hydrochlorothiazide, Quinapril

Hydrochlorothiazide, Quinapril Hydrochloride

Hydrochlorothiazide, Ramipril

Indapamide, Perindopril

Indapamide, Perindopril Erbumine

and/or 'C09BB' (ACE inhibitors and calcium channel blockers) with one of the following combination ingredients:

Trandolapril, Verapamil Hydrochloride

and/or 'C09DA' (Angiotensin II antagonists and diuretics) with one of the following combination ingredients:

Trandolapril, Verapamil Hydrochloride

Candesartan Cilexetil, Hydrochlorothiazide

Candesartan, Hydrochlorothiazide

Eprosartan Mesilate, Hydrochlorothiazide

Hydrochlorothiazide, Irbesartan

Hydrochlorothiazide, Losartan

Hydrochlorothiazide, Losartan Potassium

Hydrochlorothiazide, Olmesartan

Hydrochlorothiazide, Olmesartan Medoxomil

Hydrochlorothiazide, Telmisartan

Hydrochlorothiazide, Valsartan

and/or 'C09DX' (Angiotensin II antagonists, other combinations) with one of the following combination ingredients:

Amlodipine Besilate, Hydrochlorothiazide, Valsartan

and/or 'C09XA' (Renin-inhibitors) with one of the following combination ingredients:

Aliskiren Fumarate, Hydrochlorothiazide Aliskiren, Hydrochlorothiazide

### **ATTACHMENT 2**

Medical History and AEs of Interest Defined by MedDRA Preferred Term

#### 1. **MEDICAL HISTORY**

#### 1.1. **Hypertension**

- o Essential hypertension
- Hypertension
- o Hypertensive angiopathy
- Hypertensive cardiomyopathy
- Hypertensive crisis
- Hypertensive heart disease
- Retinopathy hypertensive

#### 1.2. **Dyslipidemia**

- Blood cholesterol
- Blood cholesterol increased
- Blood triglycerides increased
- Dyslipidaemia

- o Hypercholesterolaemia
- Hyperlipidaemia
- Hypertriglyceridaemia
- Xanthelasma

#### 1.3. **Fractures**

- Acetabulum fracture
- Hip fracture
- Ankle fracture
- Humerus fracture
- Avulsion fracture
- Ilium fracture
- o Bone fragmentation
- Impacted fracture
- o Cervical vertebral fracture
- Chance fracture
- Clavicle fracture
- Jaw fracture
- Comminuted fracture
- o Limb crushing injury
- Complicated fracture
- Lumbar vertebral fracture
- Lower limb fracture
- o Compression fracture

- Forearm fracture
- Radius fracture
- o Fracture
- o Rib fracture
- o Fracture debridement
- Scapula fracture
- o Fracture delayed union
- o Skull fracture
- o Fracture displacement
- o Skull fractured base
- o Fracture malunion
- Spinal compression
  - fracture
- o Fracture nonunion
- Sternal fracture
- o Fracture reduction
- Stress fracture
- Fractured coccyx
- Thoracic vertebral
  - fracture

- o Multiple fractures
- o Elevation skull fracture
- o Open fracture
- o Epiphyseal fracture
- Osteoporotic fracture
- o Facial bones fracture
- Patella fracture
- Femoral neck fracture
- Pathological fracture
- Femur fracture
- Pelvic fracture
- o Fibula fracture
- Pubis fracture
- Foot fracture
- o Periprosthetic fracture
- o Atypical femur fracture
- Closed fracture manipulation
- o Costal cartilage fracture
- o Craniofacial fracture
- External fixation of fracture
- o Fracture pain
- Fracture treatment
- Internal fixation of fracture
- Limb fracture
- o Loss of anatomical alignment after fracture reduction
- Open reduction of fracture
- o Open reduction of spinal fracture
- Osteochondral fracture
- Sacroiliac fracture
- Spinal fusion fracture

- o Fractured ischium
- Tibia fracture
- o Fractured sacrum
- o Torus fracture
- o Fractured maxilla elevation
- o Traumatic fracture
- Fractured skull depressed
- o Ulna fracture
- o Fractured zygomatic arch elevation
- o Upper limb fracture
- o Greenstick fracture
- o Wrist fracture
- Hand fracture
- o Spinal fracture
- Atypical fracture

## Statistical Analysis Plan 28431754DNE3001; Phase 3

# 2. LIST OF PREFERRED TERMS FOR SELECTED ADVERSE EVENTS OF INTEREST

| | Female Mycotic Genital | |
|---|---|---|
| Diabetic ketoacidosis | Infections | Fracture |
| Acidosis | Genital candidiasis | Acetabulum fracture |
| Acidosis aggravated | Genital infection | Ankle fracture |
| Acidosis diabetic | Genital infection female | Atypical femur fracture |
| Acidosis metabolic | Genital infection fungal | Atypical fracture |
| Acidosis NOS | Urogenital infection fungal | Avulsion fracture |
| Acute acidosis | Vaginal infection | Bone fragmentation |
| Anion gap acidosis | Vaginal inflammation | Cervical vertebral fracture |
| Blood ketone body | Vulvitis | Chance fracture |
| Blood ketone body increased | Vulvovaginal candidiasis | Clavicle fracture |
| | | Closed fracture manipulation |
| | | Costal cartilage fracture |
| | Vulvovaginal mycotic | |
| Blood ketone body present | infection | |
| | Vulvovaginitis | |
| | Vulvovaginal inflammation | |
| Diabetes mellitus with ketoacidosis | | Comminuted fracture |
| Diabetes with hyperosmolarity | | Complicated fracture |
| Diabetes with hyperosinolarity Diabetes with ketoacidosis | | Compression fracture |
| Diabetic acidosis | | Craniofacial fracture |
| Diabetic hyperglycemic coma | | Elevation skull fracture |
| Diabetic hyperosmolar coma | | Epiphyseal fracture |
| Diabetic hyperosmolal coma Diabetic ketoacidosis | | External fixation of fracture |
| Diabetic ketoacidosis Diabetic ketoacidotic hyperglycemic | | External fixation of fracture |
| coma | | Facial bones fracture |
| Diabetic metabolic decompensation | | Femoral neck fracture |
| High anion gap metabolic acidosis | | Femur fracture |
| Hyperglycemic seizure | | Fibula fracture |
| Hyperglycaemic hyperosmolar | | |
| nonketotic syndrome | | |
| Hyperosmolar hyperglycemic state | | Foot fracture |
| Hyperosmolar state | | Forearm fracture |
| Ketoacidosis | | Fracture |
| Ketonuria | | Fracture debridement |
| Ketosis | | Fracture delayed union |
| Metabolic acidosis | | Fracture displacement |
| Metabolic acidosis exacerbated | | Fracture malunion |
| Metabolic acidosis NOS exacerbated | | Fracture nonunion |
| Metabolic acidosis not otherwise | | |
| specified (NOS) | | Fracture pain |
| Metabolic acidosis worsened | | Fracture reduction |
| Type I diabetes mellitus with | | |
| ketoacidosis | | Fracture treatment |
| Type II diabetes mellitus with | | |
| ketoacidosis | | Fractured coccyx |
| | | Fractured ischium |
| | | Fractured maxilla elevation |
| | | Fractured sacrum |
| | | Fractured skull depressed |
| | | Fractured zygomatic arch elevation |

| | Female Mycotic Genital | |
|---|---|---|
| Diabetic ketoacidosis | Infections | Fracture |
| | | Greenstick fracture |
| | | Hand fracture |
| | | Hip fracture |
| | | Humerus fracture |
| | | Ilium fracture |
| | | Impacted fracture |
| | | Internal fixation of fracture |
| | | Jaw fracture |
| | | Limb crushing injury |
| | | Limb fracture |
| | | Loss of anatomical alignment after |
| | | fracture reduction |
| | | Lower limb fracture |
| | | Lumbar vertebral fracture |
| | | Multiple fractures |
| | | Open fracture |
| | | Open reduction of fracture |
| | | Open reduction of spinal fracture |
| | | Osteochondral fracture |
| | | Osteoporotic fracture |
| | | Patella fracture |
| | | Pathological fracture |
| | | Pelvic fracture |
| | | Periprosthetic fracture |
| | | Pubis fracture |
| | | Radius fracture |
| | | Rib fracture |
| | | Sacroiliac fracture |
| | | Scapula fracture |
| | | Skull fracture |
| | | Skull fractured base |
| | | Spinal compression fracture |
| | | Spinal fracture |
| | | Spinal fusion fracture |
| | | Sternal fracture |
| | | Stress fracture |
| | | Thoracic vertebral fracture |
| | | Tibia fracture |
| | | Torus fracture |
| | | Traumatic fracture |
| | | Ulna fracture |
| | | Upper limb fracture |
| | | Wrist fracture |

| Hepatic Injury | Hypoglycaemia | Male Mycotic Genital Infections |
|---|---|---|
| Acute graft versus host disease in liver | Hypoglycaemia | Balanitis |
| Acute hepatic failure | Hypoglycaemic coma | Balanitis candida |
| Acute yellow liver atrophy | Hypoglycaemic seizure | Balanoposthitis |
| | Blood glucose decreased | |
| Allergic hepatitis | | Balanoposthitis infective |
| | | • |

#### **Hepatic Injury** Hypoglycaemia **Male Mycotic Genital Infections** Ammonia increased Erosive balanitis Ascites Gangrenous balanitis Genital candidiasis Asterixis Autoimmune hepatitis Genital infection **Bacterascites** Genital infection fungal Biliary ascites Genital infection male Biliary cirrhosis Penile infection Biliary cirrhosis primary **Posthitis** Biliary fibrosis Bilirubin excretion disorder Biopsy liver abnormal Child-Pugh-Turcotte score increased Cholaemia Cholestasis Cholestatic liver injury Cholestatic pruritus Chronic graft versus host disease in liver Chronic hepatic failure Chronic hepatitis Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Focal nodular hyperplasia Gallbladder varices Gastric varices Gastric varices haemorrhage Graft versus host disease in liver Haemangioma of liver Haemorrhagic ascites Haemorrhagic hepatic cyst Hepatectomy Hepatic adenoma Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic cyst Hepatic cyst ruptured Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic fibrosis marker abnormal Hepatic haemangioma rupture Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic necrosis Hepatic steatosis **Hepatitis** Hepatitis acute

Hepatitis cholestatic Hepatitis chronic active

#### Hepatic Injury

#### Hypoglycaemia

**Male Mycotic Genital Infections** 

Hepatitis chronic persistent

Hepatitis fulminant

Hepatitis toxic

Hepatobiliary disease

Hepatocellular foamy cell syndrome

Hepatocellular injury

Hepatopulmonary syndrome

Hepatorenal failure

Hepatorenal syndrome

Hepatotoxicity

Hyperbilirubinaemia

Icterus index increased

Intestinal varices

Ischaemic hepatitis

Jaundice

Jaundice cholestatic

Jaundice hepatocellular

Liver and small intestine transplant

Liver disorder

Liver injury

Lupoid hepatic cirrhosis

Lupus hepatitis

Mixed liver injury

Nodular regenerative hyperplasia

Non-alcoholic steatohepatitis

Non-cirrhotic portal hypertension

Ocular icterus

Oedema due to hepatic disease

Oesophageal varices haemorrhage

Parenteral nutrition associated liver disease

Peripancreatic varices

Periportal oedema

Portal hypertension

Portal hypertensive enteropathy

Portal hypertensive gastropathy

Portal triaditis

Portal vein cavernous transformation

Portal vein dilatation

Portopulmonary hypertension

Radiation hepatitis

Renal and liver transplant

Retrograde portal vein flow

Reye's syndrome

Reynold's syndrome

Splenic varices

Splenic varices haemorrhage

Subacute hepatic failure

Varices oesophageal

Varicose veins of abdominal wall

| Malignancy Renal Cell Cancer | Malignancy Testicular | Osmotic Diuresis |
|---|---|---|
| Bladder adenocarcinoma recurrent | Apocrine breast carcinoma | Phaeochromocytoma |
| Bladder adenocarcinoma stage 0 | Breast angiosarcoma | Phaeochromocytoma crisis |
| | | Phaeochromocytoma |
| Bladder adenocarcinoma stage I | Breast angiosarcoma metastatic | excision |
| | | Phaeochromocytoma |
| Bladder adenocarcinoma stage II | Breast cancer | malignant |
| Bladder adenocarcinoma stage III | Breast cancer female | |
| Bladder adenocarcinoma stage IV | Breast cancer in situ | |
| Bladder adenocarcinoma stage unspecified | Breast cancer male | |
| Bladder cancer | Breast cancer metastatic | |
| Bladder cancer recurrent | Breast cancer recurrent | |
| Bladder cancer stage 0, with cancer in situ | Breast cancer stage I | |
| Bladder cancer stage 0, without cancer in | | |
| situ | Breast cancer stage II | |
| Bladder cancer stage I, with cancer in situ | Breast cancer stage III | |
| Bladder cancer stage I, without cancer in situ | Breast cancer stage IV | |
| Bladder cancer stage II | Breast neoplasm | |
| Bladder cancer stage III | Breast sarcoma | |
| Bladder cancer stage IV | Breast sarcoma metastatic | |
| Bladder squamous cell carcinoma recurrent | Breast sarcoma recurrent | |
| Bladder squamous cell carcinoma stage 0 | Contralateral breast cancer | |
| Bladder squamous cell carcinoma stage I | HER-2 positive breast cancer | |
| Bladder squamous cell carcinoma stage II | Hormone refractory breast cancer | |
| | Inflammatory carcinoma of breast | |
| Bladder squamous cell carcinoma stage III | recurrent | |
| | Inflammatory carcinoma of breast | |
| Bladder squamous cell carcinoma stage IV | stage III | |
| Bladder squamous cell carcinoma stage | Inflammatory carcinoma of breast | |
| unspecified | stage IV | |
| Bladder transitional cell carcinoma | Inflammatory carcinoma of the breast | |
| Bladder transitional cell carcinoma | | |
| metastatic | Intraductal papillary breast neoplasm | |
| Bladder transitional cell carcinoma recurrent | Intraductal proliferative breast lesion | |
| Bladder transitional cell carcinoma stage 0 | Invasive breast carcinoma | |
| Bladder transitional cell carcinoma stage I | Invasive ductal breast carcinoma | |
| Bladder transitional cell carcinoma stage II | Invasive lobular breast carcinoma | |
| Bladder transitional cell carcinoma stage III | Invasive papillary breast carcinoma | |
| Bladder transitional cell carcinoma stage IV | Lobular breast carcinoma in situ | |
| Metastases to bladder | Malignant nipple neoplasm | |
| Metastatic carcinoma of the bladder | Malignant nipple neoplasm female | |
| Transitional cell carcinoma | Malignant nipple neoplasm male | |

| Malignancy Renal Cell Cancer | Malignancy Testicular | Osmotic Diuresis |
|---|---|---|
| Neuroendocrine carcinoma of the bladder | | |
| | Medullary carcinoma of breast | |
| | Metaplastic breast carcinoma | |
| | Metastases to breast | |
| | Mucinous breast carcinoma | |
| | Neuroendocrine breast tumour | |
| | Nipple neoplasm | |
| | Oestrogen receptor positive breast | |
| | cancer | |
| | Paget's disease of nipple | |
| | Phyllodes tumour | |
| | Triple negative breast cancer | |
| | Tubular breast carcinoma | |
| Bladder adenocarcinoma recurrent | Apocrine breast carcinoma | Phaeochromocytoma |
| Bladder adenocarcinoma stage 0 | Breast angiosarcoma | Phaeochromocytoma crisis<br>Phaeochromocytoma |
| Bladder adenocarcinoma stage I | Breast angiosarcoma metastatic | excision |
| C | <u> </u> | Phaeochromocytoma |
| Bladder adenocarcinoma stage II | Breast cancer | malignant |
| Bladder adenocarcinoma stage III | Breast cancer female | |
| Bladder adenocarcinoma stage IV | Breast cancer in situ | |
| Bladder adenocarcinoma stage unspecified | Breast cancer male | |
| Bladder cancer | Breast cancer metastatic | |
| Bladder cancer recurrent | Breast cancer recurrent | |
| Bladder cancer stage 0, with cancer in situ | Breast cancer stage I | |
| Bladder cancer stage 0, without cancer in | | |
| situ | Breast cancer stage II | |
| Bladder cancer stage I, with cancer in situ | Breast cancer stage III | |
| Bladder cancer stage I, without cancer in situ | Breast cancer stage IV | |
| Bladder cancer stage II | Breast neoplasm | |
| Bladder cancer stage III | Breast sarcoma | |
| Bladder cancer stage IV | Breast sarcoma metastatic | |
| Bladder squamous cell carcinoma recurrent | Breast sarcoma recurrent | |
| Bladder squamous cell carcinoma stage 0<br>Bladder squamous cell carcinoma stage I | Contralateral breast cancer HER-2 positive breast cancer | |
| Bladder squamous cell carcinoma stage II | Hormone refractory breast cancer | |
| Diadder squamous cen caremonia stage ii | Inflammatory carcinoma of breast | |
| Bladder squamous cell carcinoma stage III | recurrent | |
| Bladder squamous cen caremonia stage in | Inflammatory carcinoma of breast | |
| Bladder squamous cell carcinoma stage IV | stage III | |
| Bladder squamous cell carcinoma stage | Inflammatory carcinoma of breast | |
| unspecified | stage IV | |
| 1 | Inflammatory carcinoma of the | |
| Bladder transitional cell carcinoma | breast | |
| Bladder transitional cell carcinoma | Intraductal papillary breast | |
| metastatic | neoplasm | |
| | Intraductal proliferative breast | |
| Bladder transitional cell carcinoma recurrent | lesion | |
| Bladder transitional cell carcinoma stage 0 | Invasive breast carcinoma | |
| Bladder transitional cell carcinoma stage I | Invasive ductal breast carcinoma | |
| Bladder transitional cell carcinoma stage II | Invasive lobular breast carcinoma | |
| Bladder transitional cell carcinoma stage III | Invasive papillary breast carcinoma | |

| Malignancy Renal Cell Cancer N | Malignancy Testicular | Osmotic Diuresis |
|---|---|---|
| Č | obular breast carcinoma in situ | |
| | Malignant nipple neoplasm | |
| | Malignant nipple neoplasm female | |
| | Malignant nipple neoplasm male | |
| Neuroendocrine carcinoma of the bladder | | |
| 1 | Medullary carcinoma of breast | |
| | Metaplastic breast carcinoma | |
| | Metastases to breast | |
| | Aucinous breast carcinoma | |
| N | Neuroendocrine breast tumour | |
| N | lipple neoplasm | |
| C | Destrogen receptor positive breast | |
| | ancer | |
| | aget's disease of nipple | |
| | hyllodes tumour | |
| | riple negative breast cancer Subular breast carcinoma | |
| | Benign neoplasm of testis | Dry mouth |
| | Leydig cell tumour of the testis | Dry throat |
| | Sertoli cell testicular tumour | Micturition disorder |
| Hereditary leiomyomatosis renal cell | | |
| | Spermatocytic seminoma | Micturition urgency |
| J I II | Testicle adenoma | Nocturia |
| | Testicular cancer metastatic | Pollakiuria |
| * | Festicular neoplasm | Polydipsia |
| · | Гesticular papilloma<br>Гestis cancer | Polyuria<br>Thirst |
| Renal cancer metastatic | resus cancer | Tongue dry |
| Renar cancer metastatic | | Urine output |
| Renal cancer recurrent | | increased |
| Renal cancer stage I | | |
| Renal cancer stage II | | |
| Renal cancer stage III | | |
| Renal cancer stage IV | | |
| Renal cell carcinoma | | |
| Renal cell carcinoma recurrent | | |
| Renal cell carcinoma stage I<br>Renal cell carcinoma stage II | | |
| Renal cell carcinoma stage II | | |
| Renal cell carcinoma stage IV | | |
| Rhabdoid tumour of the kidney | | |
| Papillary renal cell carcinoma | | |

| Phimosis | Photosensitivity |
|-------------------|-----------------------------------------------|
| Acquired phimosis | Actinic elastosis |
| Phimosis | Actinic prurigo |
| | Administration site photosensitivity reaction |
| | Application site photosensitivity reaction |
| | Chronic actinic dermatitis |
| | Hartnup disease |
| | Implant site photosensitivity |
| | Infusion site photosensitivity reaction |
| | Injection site photosensitivity reaction |
| | Juvenile spring eruption |
| | Medical device site photosensitivity reaction |
| | Photodermatosis |
| | Photokeratitis |
| | Photoonycholysis |
| | Photosensitivity reaction |
| | Polymorphic light eruption |
| | Solar dermatitis |
| | Solar urticaria |
| | Sunburn |
| | Vaccination site photosensitivity reaction |

| Renal Related | Severe Hypersensitivity/Cutaneous AEs | Upper UTI |
|---|---|---|
| Acute kidney injury | Acute generalised exanthematous pustulosis | Bacterial pyelonephritis |
| | | Emphysematous |
| Acute phosphate nephropathy | Allergic oedema | pyelonephritis |
| Acute prerenal failure | Anaphylactic reaction | Kidney infection |
| Anuria | Anaphylactic shock | Perinephric abscess |
| Azotaemia | Anaphylactic transfusion reaction | Pyelocystitis |
| Blood creatinine increased | Anaphylactoid reaction | Pyelonephritis |
| Blood urea increased | Anaphylactoid shock | Pyelonephritis acute |
| Continuous | • • | • |
| haemodiafiltration | Angioedema | Pyelonephritis chronic |
| Dialysis | Circulatory collapse | Pyelonephritis fungal |
| Glomerular filtration rate | • | Pyelonephritis |
| decreased | Circumoral oedema | mycoplasmal |
| Haemodialysis | Conjunctival oedema | Pyelonephritis viral |
| Haemofiltration | Corneal exfoliation | Pyonephrosis |
| Hypercreatininaemia | Corneal oedema | Renal abscess |
| Neonatal anuria | Cutaneous vasculitis | Renal cyst infection |
| Nephritis | Dermatitis bullous | Urosepsis |
| | | Pyelitis |
| Nephropathy toxic | Dermatitis exfoliative | |
| Oliguria | Dermatitis exfoliative generalised | |
| Peritoneal dialysis | Drug eruption | |
| Prerenal failure | Drug hypersensitivity | |
| | Drug reaction with eosinophilia and systemic | |
| Renal failure | symptoms | |
| Renal failure acute | Epidermal necrosis | |
| Renal failure neonatal | Epiglottic oedema | |
| Renal impairment | Erythema multiforme | |
| Renal impairment neonatal | Exfoliative rash | |
| | Eye oedema | |
| | Eye swelling | |
| | | 48 |

## **Renal Related** Severe Hypersensitivity/Cutaneous AEs **Upper UTI** Eyelid oedema Face oedema First use syndrome Fixed drug eruption Gingival oedema Gingival swelling Gleich's syndrome Hereditary angioedema Hypersensitivity vasculitis Idiopathic angioedema Idiopathic urticaria Kounis syndrome Laryngeal dyspnoea Laryngeal oedema Laryngospasm Laryngotracheal oedema Limbal swelling Lip exfoliation Lip oedema Lip swelling Mucocutaneous ulceration Mucosa vesicle Mucosal erosion Mucosal exfoliation Mucosal necrosis Mucosal ulceration Nikolsky's sign Oculomucocutaneous syndrome Oculorespiratory syndrome Oedema mouth Oedema mucosal Oral mucosal blistering Oral mucosal exfoliation Orbital oedema Oropharyngeal blistering Oropharyngeal swelling Palatal oedema Penile exfoliation Periorbital oedema Pharyngeal oedema Scleral oedema Shock Shock symptom Skin exfoliation Skin necrosis Small bowel angioedema Stevens-Johnson syndrome Stridor Swelling face Swollen tongue Symmetrical drug-related intertriginous and flexural exanthema Throat tightness Tongue exfoliation

| Renal Related | Severe Hypersensitivity/Cutaneous AEs | Upper UTI |
|---------------|---------------------------------------|-----------|
| | Tongue oedema | |
| | Toxic epidermal necrolysis | |
| | Type I hypersensitivity | |
| | Urticaria | |
| | Urticaria cholinergic | |
| | Urticaria chronic | |
| | Urticaria papular | |
| | Urticarial vasculitis | |
| | Vaginal exfoliation | |

| UTI | Venous Thromboembolic events | Volume Depletion |
|---|---|---|
| Bacterial ureteritis | | • |
| Bacterial urethritis | | |
| Bladder candidiasis | Deep vein thrombosis | Blood pressure decreased |
| Cystitis | Deep vein thrombosis postoperative | Blood pressure orthostatic decreased |
| Cystitis bacterial | Embolism venous | Dehydration |
| Cystitis escherichia | Iliac vein occlusion | Diastolic hypotension |
| Cystitis gonococcal | Inferior vena cava syndrome | Dizziness postural |
| Cystitis haemorrhagic | Inferior vena caval occlusion | Hypotension |
| Cystitis interstitial | Jugular vein occlusion | Hypovolaemia |
| Cystitis klebsiella | Mesenteric venous occlusion | Hypovolaemic shock |
| Cystitis pseudomonal | Obstructive shock | Orthostatic hypotension |
| • | Portosplenomesenteric venous | |
| Emphysematous cystitis | thrombosis | Orthostatic intolerance |
| | | Postural orthostatic tachycardia |
| Escherichia urinary tract infection | Post procedural pulmonary embolism | syndrome |
| Fungal cystitis | Postpartum venous thrombosis | Presyncope |
| Funguria | Pulmonary embolism | Shock |
| Genitourinary tract infection | Pulmonary infarction | Shock symptom |
| Streptococcal urinary tract | | |
| infection | Pulmonary microemboli | Syncope |
| Ureter abscess | Pulmonary oil microembolism | Urine output decreased |
| Ureteritis | | |
| Urethritis | | |
| Urethritis noninfective | Pulmonary thrombosis | |
| Uretheritis | Renal vein embolism | |
| Urethral abscess | Renal vein occlusion | |
| Urethral carbuncle | Subclavian vein thrombosis | |
| Urethral stricture post infection | Vascular occlusion | |
| Urinary bladder abscess | Venous thrombosis | |
| Urinary tract abscess | Venous thrombosis in pregnancy | |
| Urinary tract infection | Venous thrombosis limb | |
| Urinary tract infection bacterial | Visceral venous thrombosis | |
| Urinary tract infection | | |
| enterococcal | | |
| Urinary tract infection fungal | | |
| Urinary tract infection | | |
| pseudomonal | | |
| Urinary tract infection | | |
| staphylococcal | | |

### **ATTACHMENT 3**

## **CLINICAL LABORATORY TESTS**

The clinical laboratory tests include following panels and assessments:

- Hematology panel
  - o hemoglobin
  - o platelet count
  - o hematocrit
  - o red blood cell (RBC) count
  - o white blood cell (WBC) count with differential
- Serum chemistry panel
  - o Sodium
  - potassium
  - chloride
  - bicarbonate
  - BUN 0
  - o creatinine
  - o aspartate aminotransferase (AST)
  - alanine aminotransferase (ALT)

  - gamma-glutamyltransferase (GGT)
  - total bilirubin

- o alkaline phosphatase
- creatine phosphokinase (CPK)
- lactic acid dehydrogenase (LDH)
- uric acid 0
- calcium 0
- phosphate
- albumin 0
- total protein 0
- magnesium

- Urinalysis
- Lipid panel
  - Triglycerides
  - o Total cholesterol
  - HDL cholesterol
  - o LDL cholesterol
  - LDL/HDL ratio
- Plasma glucose
- Hemoglobin A<sub>1c</sub>
- **Estimated Glomerular Filtration Rate (eGFR)**

The estimated glomerular filtration rate (eGFR) will be reported according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at study visits when serum creatinine is measured by the central laboratory.

## **ATTACHMENT 4**

# CRITERIA FOR PRE-DEFINED LIMIT OF CHANGE (PDLC) AND ABNORMAL VALUES

| Laboratory Test | Parameter for ANY value and LAST value |
|---|---|
| CHEMISTRY | |
| | Absolute Value: >3X ULN |
| ALT | Absolute Value: >5X ULN |
| | Absolute Value: >8X ULN |
| | Absolute Value: >3X ULN |
| AST | Absolute Value: >5X ULN |
| | Absolute Value: >8X ULN |
| | Composite: ALT >3X ULN and Tbili >2X ULN [with the Tbili elevation >2 X |
| ALT >3X ULN and Tbili >2X ULN | ULN within 30 days of the ALT elevation >3x ULN] |
| | Composite: AST >3X ULN and Tbili >2X ULN [with the Tbili elevation >2 X |
| AST >3X ULN and Tbili >2X ULN | ULN within 30 days of the AST elevation >3x ULN] |
| | Composite: >ULN and > 25% increase from BL |
| Bilirubin | Absolute Value: >2XULN |
| Bicarbonate | Absolute Value: <16 mEq/L |
| Calcium | Composite: >ULN and > 10 % increase from BL |
| eGFR from creatinine adjusted for | eGFR < 80 mL/min/1.73m2 and decrease > 30% from BL |
| BSA | eGFR decrease > 50% from BL |
| | Composite: <lln and="">25% decrease from BL</lln> |
| Magnesium | Composite: >ULN and >25% increase from BL |
| _ | Composite: <lln and="">25% decrease from BL</lln> |
| Phosphate | Composite: >ULN and >25% increase from BL |
| | Composite: <lln and="">15% decrease from BL</lln> |
| Potassium | Composite: >ULN and >15% increase from BL |
| | Absolute Value: ≥ 6.5 mEq/L |
| | Composite: <lln and="" decrease="">5 mEq/L or more from BL</lln> |
| Sodium | Composite: >ULN and increase>5 mEq/L or more from BL |
| Albumin | Composite: <lln and="">25% decrease from BL</lln> |
| Urate | Composite: <lln and="">25% decrease from BL</lln> |
| HEMATOLOGY | |
| | Change: ≥ 2 g/dl decrease from BL |
| Hemoglobin | Change: ≥ 2 g/dL increase from BL |
| Platelets | Composite: <lln and="" decrease="">25% from BL</lln> |
| | Composite: >ULN and increase >25% from BL |
| | Composite: < LLN and >25% decrease from BL |
| White Blood Count | Composite: > ULN and >50 % increase from BL |
| VITAL SIGNS | |
| | Absolute Value: ≤50 beats per minute |
| Pulse | Absolute Value: ≥100 beats per minute |
| | Composite: ≥ 20 mm Hg decrease from BL and ≤90 mm Hg |
| Systolic Blood Pressure | Composite: ≥ 20 mm Hg increase from BL and ≥ 160 mm Hg |
| | Composite: ≥ 15 mm Hg decrease from BL and ≤ 50 mm Hg |
| Diastolic Blood Pressure | Composite: ≥ 15 mm Hg increase from BL and ≥ 100 mm Hg |